CLINICAL TRIAL: NCT05006521
Title: Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, PK, and PD of Single Ascending Doses of KN-002 in Healthy Subjects and Multiple Ascending Doses of KN-002 in Subjects With Mild Asthma, Moderate-Severe Asthma and COPD
Brief Title: Single and Multiple Ascending Dose Study of KN-002
Acronym: KN-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinaset Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KN-002/1/001
Record Dates: First submitted 2021-07-30; First posted 2021-08-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Asthma COPD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- KN-002 for SAD (Part 1) (Experimental): Up to 6 cohorts with 6 of 8 subjects per cohort randomised to receive KN-002
  Interventions: Drug: KN-002
- Placebo for SAD (Part 1) (Placebo Comparator): Up to 6 cohorts with 2 of 8 subjects per cohort randomised to receive placebo
  Interventions: Drug: KN-002
- KN-002 for MAD (Part 2) (Experimental): Up to 4 cohorts with 6 of 8 subjects per cohort randomised to receive KN-002
  Interventions: Drug: KN-002
- Placebo for MAD (Part 2) (Experimental): Up to 4 cohorts with 2 of 8 subjects per cohort randomised to receive placebo
  Interventions: Drug: KN-002
- KN-002 for Part 3 (Experimental): Single cohort with up to 18 of 24 subjects randomised to active treatment
  Interventions: Drug: KN-002
- Placebo for Part 3 (Experimental): Single cohort with up to 6 of 24 subjects randomised to placebo treatment
  Interventions: Drug: KN-002
- KN-002 for Part 4 (Experimental): Single cohort with up to 18 of 24 subjects randomised to active treatment
  Interventions: Drug: KN-002
- Placebo for Part 4 (Experimental): Single cohort with up to 6 of 24 subjects randomised to placebo treatment
  Interventions: Drug: KN-002

INTERVENTIONS:
Drug: KN-002 — KN-002 dry powder inhaler

SUMMARY:
This is a Phase 1, randomized, double-blinded, placebo controlled study. The study consists of 4 parts: Part 1 is a single ascending dose (SAD) study in healthy volunteers; Part 2 is a multiple ascending dose (MAD) study in subjects with stable, mild asthma; Part 3 is a repeat dose in patients with moderate to severe asthma and Part 4 is a repeat dose in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 55 years old
* Willing and able to give informed consent and comply with the study
* Body mass index (BMI) 18 to 32 kg/m2 and weighs at least 50 kg
* Women of child bearing potential must have a negative pregnancy test and use a highly efficient birth control method
* Pre-bronchodilator FEV1 ≥ 70 and ≥80% for Part 1 and Part 2 participants, respectively
* Pre-Bronchodilator FEV1 ≥50% predicted and ≤100% for Part 3
* Post Bronchodilator FEV1 ≥40 and ≤ 85% for Part 4

Exclusion Criteria:

* Clinically significant laboratory test abnormalities
* Clinically significant abnormal blood pressure and/or pulse rate
* Resting ECG clinically significant abnormalities
* Respiratory tract infection within 6 weeks of screening
* Positive test for active COVID-19 within 2 days prior to administration of IMP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Parts 1, 2, 3 and 4) via an assessment of the incidence of treatment-related adverse events | Day 1 to 17
  To assess the safety and tolerability of KN-002 via the assessment of the number, severity and type of treatment emergent adverse events post single and repeat dose administration to healthy volunteers and patients with mild asthma, moderate to severe asthma and COPD

SECONDARY OUTCOMES:
Pharmacokinetics (Parts 1, 2, 3 and 4) via the determination of area under the curve (AUC) | Day 1 to 17
  KN-002 pharmacokinetics after single and repeat dosing to healthy volunteers and patients with mild asthma, moderate to severe asthma and COPD:
Pharmacokinetics (Parts 1, 2, 3 and 4) via the determination of maximum plasma concentrations (Cmax) | Day 1 to 17
  KN-002 pharmacokinetics after single and repeat dosing to healthy volunteers and patients with mild asthma, moderate to severe asthma and COPD:
Pharmacodynamics (Parts 2, 3 and 4) via changes in fractional exhaled nitric oxide (FeNO) levels | Day 1 to 17
  Change of fractional exhaled nitric oxide (FeNO) levels after repeated dosing to patients with mild asthma, moderate to severe asthma and COPD

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicines Evaluation Unit
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Kinaset Therapeutics Inc. will not disclose individual subject de-identified study data